CLINICAL TRIAL: NCT02460601
Title: The Efficacy and Safety of Qizhiweitong Granule on Patients With Functional Dyspepsia in a Multi-center Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhongcheng Duan, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCMSBL-09006
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Qizhiweitong granule (Experimental): 2.5g/time,tid,oral administration,6 weeks
  Interventions: Drug: Qizhiweitong granule
- Placebo (Placebo Comparator): 2.5g/time,tid,oral administration,6 weeks
  Interventions: Drug: Qizhiweitong granule

INTERVENTIONS:
Drug: Qizhiweitong granule

SUMMARY:
The study aims to verify the efficacy and safety of Qizhiweitong granule on Chinese patients with functional dyspepsia diagnosed by the Rome III criteria. It includes two subtypes of functional dyspepsia, postprandial distress syndrome or abdominal pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. patient with written ICF signed
2. patient with functional dyspepsia diagnosed by the Rome III criteria
3. age between 18y and 65y;male or female.
4. patient without gastric ulcers, erosive gastritis or other gastric organic diseases according to the endoscopy in the past one year in the hospital
5. patient without hepatobiliary and pancreatic diseases according to B-ultrasoundin the past one year in the hospital
6. patient with normal ECG (QT interval in the normal range) within one month prior to enrollment in this center
7. patient with symptoms of only one subtype of functional dyspepsia

Exclusion Criteria:

1. history of abdominal surgery;
2. take drugs related to gastrointestinal motility or gastric acid secretion and gastric acid drugs, anti-Helicobacter pylori drugs within 5 days of inclusion
3. suffering from hepatobiliary and pancreatic diseases with B ultrasound
4. suffering from high blood pressure and uncontroled hypertension
5. diabetes mellitus
6. have history of thyroid disease, systemic sclerosis, systemic lupus erythematosus
7. severe mental disorders
8. pregnant women, breastfeeding women or those who plan to become pregnant
9. allergy to Qizhiweitong particle
10. have symptoms of both subtypes of functional dyspepsia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
symptom severity score | 3 days

REFERENCES:
- [Derived] Su Q, Chen SL, Wang HH, Liang LX, Dai N, Lyu B, Zhang J, Wang RQ, Zhang YL, Yu Y, Liu JS, Hou XH. A Randomized, Double-Blind, Multicenter, Placebo-Controlled Trial of Qi-Zhi-Wei-Tong Granules on Postprandial Distress Syndrome-Predominant Functional Dyspepsia. Chin Med J (Engl). 2018 Jul 5;131(13):1549-1556. doi: 10.4103/0366-6999.235118. PMID 29941708